CLINICAL TRIAL: NCT06284265
Title: Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Clinical Trial of the Efficacy and Safety of Raphamin in Prevention of the Recurrences of Chronic Bacterial Cystitis
Brief Title: Clinical Trial of the Efficacy and Safety of Raphamin in Prevention of Recurrences of Chronic Bacterial Cystitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMH-407-007
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cystitis Chronic; Cystitis Bacterial; Recurrence of Chronic Bacterial Cystitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raphamin (Experimental): Take orally, do not take with meals. Keep the tablets in the mouth until completely dissolved.
  On the first day of treatment, 8 tablets are taken according to the following scheme: 1 tablet every 30 minutes in the first 2 hours (a total of 5 tablets in 2 hours), then during the same day another 1 tablet is taken 3 times at regular intervals. On the 2nd day and then take 1 tablet 3 times a day. The duration of treatment is 10 days.
  Interventions: Drug: Raphamin
- Placebo (Placebo Comparator): Take orally, do not take with meals. Keep the tablets in the mouth until completely dissolved. Placebo is administered according to the Raphamin regimen for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raphamin — Tablet for oral use.
  Other Names: MMH-407
  Arms: Raphamin
Drug: Placebo — Tablet for oral use.
  Arms: Placebo

SUMMARY:
Clinical Trial of the Efficacy and Safety of Raphamin in Prevention of Recurrences of Chronic Bacterial Cystitis

DETAILED DESCRIPTION:
Trial design: double blind, placebo-controlled, randomized in parallel groups clinical trial.

The trial includes female outpatients aged 18 years or older with typical symptoms of chronic bacterial cystitis. The severity of typical symptoms of recurrence (exacerbation) should be 7 points or more according to the subscale "Typical symptoms" of the scale "Acute Cystitis Symptom Scale" (ACSS).

At Visit 1 (Day 1), after signing the patient information sheet and the informed consent form for participation in the clinical trial, complaints and medical history are collected, a physical examination is performed, and the severity of typical symptoms of cystitis is assessed using ACSS, collection of urine biosamples for urine analysis with microscopy and bacteriological examination (for identification the sensitivity of microorganisms to antibiotics), ultrasound examination of the urinary system (kidneys, bladder), and concomitant therapy is recorded.

Urinalysis, general and biochemical blood tests are planned in at least 190 patients.

If the patient meets inclusion criteria and does not meets exclusion inclusion criteria at Visit 1 (Day 1), the patient is randomized to one of two groups: patients of Group 1 take Phosphomycin (3 g once) and Raphamin according to the therapeutic and preventive regimen for 10 days; patients of Group 2 use Phosphomycin (3 g once) and Placebo according to the Raphamin regimen for 10 days.

If there is no effect from treatment within 48 hours or phosphomycin-resistant strains are detected, the physician conducts unscheduled visit and gives the patient an alternative drug Cefixime (400 mg). Cefixime is taken 1 times a day at a dose of 400 mg for 5 days or more (the duration of the course is determined by the physician).

All patients are provided with Phosphomycin, if resistance to it is detected - with alternative antibiotic Cefixime.

If microorganisms resistant to both Phosphomycin and Cefixime are detected, the patient is excluded from the trial, and the physician prescribes a treatment strategy in accordance with current standards.

In Electronic Patient Diary (EPD) the patient records the severity of typical cystitis symptoms using ACSS once a day at approximately the same time. Symptoms are recorded in the EPD from the patient's enrollment until Visit 2 (within 10 days of study drug administration), as well as during 10 days of treatment for each subsequent relapse (exacerbation).

In addition, any possible deterioration of the patient's condition (if applicable) is recorded in EDP to assess safety and record adverse events. The study physician instructs patients to complete the diary.

The first ACSS marks in the EDP are made by patient together with physician at Visit 1. EDP is available for filling throughout the patient's participation in the study. Once a week, the patients get SMS reminder: "If you have symptoms of the disease, enter them in the diary and contact the study physician. Don't forget to take your medication." In total, patient's follow-up lasts for 24 weeks. In the process of treatment and observation, 4 visits are scheduled: at day 1 (Visit 1) and day 11 (Visit 2), then at weeks 12 and 24 (Visits 3, 4). Visits 1, 2 and 4 are face-to-face (patient visits trial site); physician conducts physical examination, records symptoms and concomitant therapy, and checks the EPD. At Visit 2 (Day 11+3), the physician gives Phosphomycin/Cefixime and a study drug to patient, to treat a possible subsequent recurrence of cystitis. Blood and urine biosamples are taken from the patient who signed the ICF for taking biological samples (for safety assessment). The study drug received by the patient at Visit 1 should be returned to assess the patient's adherence to the study treatment. Phosphomycin/Cefixime also returns.

Visit 3 (Week 12 ± 3 days) is conducted by correspondence (telephone), in order to interview the patient about her condition.

In case of new recurrence of cystitis, patient contacts with trial physician by phone. On the basis of complaints and symptoms, physician makes conclusion about the onset of chronic cystitis recurrence. Patient completes ACSS in EPD. For a recurrence of cystitis, patient takes Phosphomycin (or Cefixime) and trial product (Raphamin/Placebo for 10 days). At the end of 10 days of treatment, an unscheduled face-to-face visit takes place (Day 11+3 days after the onset of recurrence), at which the patient returns the trial product and Phosphomycin/Cefixime, then the physician dispenses a new pack of trial product and Phosphomycin (or Cefixime) to treat a possible new recurrence of cystitis.

Visit 4 (Week 24 ± 3 days) is the final one; complaints are assessed, the patient undergoes a physical examination, returns the trial product and fills in a visual analogue scale (VAS), which assesses the degree of patient satisfaction with the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 years and older.
2. Patients with a confirmed diagnosis of chronic bacterial cystitis.
3. Patients with exacerbation of chronic cystitis based on typical symptoms of exacerbation of the disease with a severity of 7 points or more in accordance wuth ACSS.
4. The first 48 hours from the onset of exacerbation) of chronic bacterial cystitis.
5. Patients who agreed to use an acceptable method of contraception during the study (for women of reproductive potential).
6. Availability of a signed patient information sheet and informed consent form for participation in the clinical trial.

Exclusion Criteria:

1. Presence of urolithiasis, urinary tract obstruction, urothelial cancer, pelvic organ prolapse, neurogenic bladder disorders at the time of examination.
2. Presence of malignant neoplasms of the urinary tract, ureter stone, more than 50 ml of residual urine in the bladder, confirmed by ultrasound examination.
3. Suspicion of bladder tuberculosis.
4. Presence of indications for hospitalization due to a serious condition, macrohematuria, complicated cystitis.
5. Decompensation of diabetes mellitus, immunodeficiency of any etiology, malignant cancer of any localization, severe circulatory insufficiency (cardiovascular disease with functional class IV according to the classification of the New York Heart Association, 1964).
6. Unstable angina pectoris or myocardial infarction within the previous 6 months.
7. Chronic kidney disease (classes С3-5 А3).
8. Hepatic impairment (Child-Pugh class C).
9. Patients who require medicinal products prohibited for use in this study.
10. Exacerbation or decompensation of chronic conditions affecting the patient's ability to participate in the clinical trial.
11. Malabsorption syndrome, including congenital or acquired lactase deficiency or other disaccharidase insufficiency, galactosemia.
12. Hypersensitivity to any component of the medicinal products used in the treatment.
13. Pregnancy, breastfeeding; childbirth less than 3 months prior to study enrollment, unwillingness to comply with contraceptive methods during the study.
14. The medications listed in the Prohibited Concomitant Medication section were administered within 4 weeks prior to enrollment.
15. Patients who, from the investigator's point of view, will not comply with the observation requirements of the study or comply with the administration of the study drug.
16. History of mental diseases, alcoholism, or drug abuse that, in the investigator's opinion, may interfere with the successful completion of trial procedures.
17. Participation in other clinical trials within 3 months prior to enrollment.
18. The patient belongs to the investigational site personnel directly involved in the study, closest relatives of the investigator. The closest relatives are defined as spouse, parents, children or siblings, regardless of whether they are natural or adopted.
19. The patient works for the company OOO "NPF "MATERIA MEDICA HOLDING", being an employee of the company, a temporary contract worker or an appointed official responsible for performing the trial, or their close relative.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to the first recurrence of chronic bacterial cystitis | 6 months
  Criteria for the diagnosis of chronic bacterial cystitis recurrence are typical symptoms of exacerbation (acute cystitis): frequent urination with small volumes of urine; urgent urination (a sudden and uncontrollable urge to pass urine; feeling pain or burning when passing urine; feeling of incomplete bladder emptying after urination; pain or uncomfortable pressure in the lower abdomen (above the pubis); possible presence of blood in the urine (especially towards the end of urination).
  Criteria for the diagnosis of chronic bacterial cystitis are 2 and more recurrences during previous 6 months or 3 and more recurrences during previous 12 months.

SECONDARY OUTCOMES:
Percentage of patients with a reduction of recurrences of chronic bacterial cystitis | 6 months
  Percentage of patients with a reduction number of recurrences of chronic bacterial cystitis to one episode and less during 6 months of follow-up.

OTHER OUTCOMES:
Average duration of episodes of recurrences of chronic bacterial cystitis | 6 months
  Average duration of episodes of recurrences of chronic bacterial cystitis after the start of study therapy at inclusion in the study, score 6 or less of typical symptoms of cystitis by the Acute Cystitis Symptom Score (according to the patient's diary).
Average number of recurrences of chronic bacterial cystitis | 6 months
  Average number of recurrences of chronic bacterial cystitis per patient during 6 months of follow-up.
Severity of chronic bacterial cystitis recurrences | 6 months
  Severity of chronic bacterial cystitis recurrences within 6 months of follow-up (as measured by the area under the curve for the total score of typical symptoms of cystitis on the Acute Cystitis Symptom Score (ACSS) during 10 days of treatment for each episode of recurrence).
  ACSS is an 18-item self-reporting questionnaire for clinical diagnosis and follow-up of acute uncomplicated cystitis in women (min 0, max 18 points; 6 typical symptoms are included: urinary frequency, urgent urination, burning feeling when urinating, incomplete bladder empting after urination, pain or uncomfortable pressure in the lower abdomen, visible blood in urine; each symptom is estimated from 0 to 3 points).
Change in the severity of chronic bacterial cystitis recurrences | 6 months
  Change in the severity of chronic bacterial cystitis recurrences during 6 months of follow-up compared to baseline.
VAS score at the end of the follow-up period | 6 months
  Visual Analogue Scale (VAS) is used to assess the degree of satisfaction with the treatment. Treatment satisfaction scores are ranged from 0 (no satisfaction with treatment) to 10 points (very significant treatment effect), such that a higher score indicates greater treatment efficacy.
The Presence of Adverse Events (AEs). | 6 months
  The presence and nature of adverse events, their intensity (severity), causal relationship to the study drug, outcome. Based on medical records.
Changes in Vital Signs (Blood Pressure measured in mm Hg) | 6 months
  Changes in Blood Pressure at the end of treatment of the initial recurrence of chronic cystitis.
Changes in Vital Signs (Pulse Rate (Heart Rate) measured in beats per minute) | 6 months
  Changes in Heart Rate at the end of treatment of the initial recurrence of chronic cystitis.
Changes in Vital Signs (Respiration Rate (Breathing Rate) measured in breaths per minute) | 6 months
  Changes in Respiratory Rate at the end of treatment of the initial recurrence of chronic cystitis.
  Based on medical records.
Proportion of patients with clinically significant laboratory abnormalities | 6 months
  Proportion of patients with clinically significant laboratory findings abnormalities at the end of treatment for initial recurrence of chronic cystitis.

CONTACTS AND LOCATIONS:
Locations (57):
- Russia (57):
  - Scientific Center for Family Health and Human Reproduction Problems/Reproductive Health Department, Irkutsk
  - Kazan State Medical University/Professor's clinic, Kazan'
  - LLC "Fenareta" Women's and Men's Health Clinic", Kemerovo
  - City Clinical Hospital #15 named after O.M. Filatov Department of Health of Moscow, Moscow
  - City Clinical Hospital # 13/Gynecology Department # 1, Moscow
  - Clinical Hospital # 85 of the Federal Medical and Biological Agency/Central polyclinic, Moscow
  - Research Institute of Rheumatology named after V.A. Nasonova, Moscow
  - National Medical Research Center for Obstetrics, Gynecology and Perinatology named after V.I. Kulakov/Department of Aesthetic Gynecology and Rehabilitation, Moscow
  - Peoples' Friendship University of Russia/Department of Obstetrics and Gynecology with a course in perinatology, Moscow
  - Russian National Research Medical University named after N.I. Pirogov/Department of Obstetrics and Gynecology, Faculty of Medicine, Moscow
  - City Clinical Hospital # 1 named after. N.I. Pirogov of the Moscow City Health Department, Moscow
  - United hospital with clinic of the Administration of the President of the Russian Federation, Moscow
  - City Clinical Hospital # 67 named after L.A. Vorokhobov, Moscow
  - JSC "MEDSI Group of Companies", Moscow
  - Moscow State Medical and Dental University named after A.I. Evdokimov/Department of Urologya, Moscow
  - Privolzhsky District Medical Center, Nizhny Novgorod
  - National Medical Research Center for Radiology/Research Institute of Urology and Interventional Radiology named after. N.A. Lopatkin, Obninsk
  - LLC "Urology Clinic # 1", Penza
  - City Clinical Hospital, Pyatigorsk
  - Rostov Central District Hospital, Rostov
  - Clinical and Diagnostic Center "Health" in Rostov-on-Don, Rostov-on-Don
  - Rostov State Medical University/Department of Urology and Human Reproductive Health with a course of pediatric urology-andrology, Rostov-on-Don
  - Ryazan State Medical University named after Academician I.P. Pavlov/Department of Urology with a course of surgical diseases, Ryazan
  - JSC "Polyclinic Complex", Saint Petersburg
  - LLC "Medical Center Capital-Polis", Saint Petersburg
  - City Geriatric Medical and Social Center, Saint Petersburg
  - LLC "BioTechService", Saint Petersburg
  - City clinic # 44, Saint Petersburg
  - All-Russian Center for Emergency and Radiation Medicine named after A.M. Nikiforov/Urology department, Saint Petersburg
  - St. Luke's Clinical Hospital, Saint Petersburg
  - City Multidisciplinary Hospital # 2/Urology department, Saint Petersburg
  - Llc "Medical Clinic", Saint Petersburg
  - Medical and sanitary unit No. 70 - branch of the St. Petersburg State Unitary Enterprise of Passenger Road Transport, Saint Petersburg
  - City Polyclinic # 112, Saint Petersburg
  - LLC "Research Center Eco-Safety", Saint Petersburg
  - Jsc "Northwestern Center of Evidence-Based Medicine", Saint Petersburg
  - LLC "Zvezdnaya Clinic", Saint Petersburg
  - City Hospital # 33, Saint Petersburg
  - LLC "New clinic "ABIA", Saint Petersburg
  - LLC "Medical Center "PRIME ROSE", Saint Petersburg
  - City Hospital # 15, Saint Petersburg
  - Research Institute of Obstetrics, Gynecology and Reproductology named after D.O. Ott/Department of Gynecology and Endocrinology, Saint Petersburg
  - City Pokrovskaya Hospital/Department of Urology, Saint Petersburg
  - City Polyclinic # 3, Saint Petersburg
  - City Polyclinic # 4, Saint Petersburg
  - LLC "Health Formula", Semiluki
  - Sertolovo City Hospital, Sertolovo
  - LLC "Uromed", Smolensk
  - Siberian State Medical University/Faculty clinics of Siberian State Medical University, Tomsk
  - Tver State Medical University/Department of Obstetrics and Gynecology, Tver'
  - Bashkir State Medical University/Department of Obstetrics and Gynecology # 1, Ufa
  - Voronezh State Medical University named after N.N. Burdenko/Department of Urology, Voronezh
  - Vsevolozhsk Clinical Interdistrict Hospital/Center for Outpatient Surgery, Vsevolozhsk
  - Yaroslavl State Medical University/Department of Urology and Nephrology, Yaroslavl
  - LLC "Clinic of Modern Medicine Dr. Bogorodskaya", Yaroslavl
  - LLC "Medical Center for Diagnosis and Prevention Plus", Yaroslavl
  - Regional Clinical Hospital/Urology department, Yaroslavl